CLINICAL TRIAL: NCT05007600
Title: Investigating the Effectiveness of Online Interactive Courses on Loneliness and Quality of Life of Older Adults in the Community During COVID-19 Pandemic: A Pilot Study and a Randomized Controlled Trial
Brief Title: Online Interactive Courses on Loneliness and Quality of Life of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Shang-Yu (Other)
Responsible Party: Sponsor-Investigator, Yang Shang-Yu, Assistant professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CRREC-109-088
Record Dates: First submitted 2021-08-05; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Older Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): Participants in the experimental group received an 8-week intensive (Monday to Friday) online interactive course.
  Interventions: Other: Online Interactive Courses
- Control group (No Intervention): Participants in the control group consumed 8 weeks of unidirectional online video and audio programs (such as from YouTube).

INTERVENTIONS:
Other: Online Interactive Courses — In the experimental group, after consensus was reached in the expert meeting (consisting of a doctor specializing in occupational therapy, a doctor specializing in nursing, and a doctor specializing in public health), a 5-days-per-week (Monday to Friday) 8-week intensive online interactive course was designed. The course was made accessible to the participants through a social network app (Line) from 12:00 to 20:30.
  Arms: trial group

SUMMARY:
Background:

The early stage of the COVID-19 pandemic can be marked as a critical period in human history as it increased loneliness in people's lives. This is particularly true for the older adults who are single, living alone, and suffering from chronic diseases. However, there is insufficient existing research on associated interventions and their effectiveness.

Objectives:

To investigate the effectiveness of an 8-week online interactive course on the loneliness, depression, social support, and quality of life (QOL) of older adults in the community during the COVID-19 pandemic.

Methods:

This pilot study, also a single-blind randomized controlled trial, collected data from a community in central Taiwan. Participants were randomly divided into an experimental group and a control group. Subsequently, participants in the experimental group received an 8-week intensive (Monday to Friday) online interactive course, whereas those in the control group consumed 8 weeks of unidirectional online video and audio programs (such as from YouTube). Assessments were conducted both before and after the intervention, with the primary outcome being the UCLA Loneliness Scale (UCLA), and secondary outcomes being the Geriatric Depression Scale Short Form, the Inventory of Socially Supportive Behavior (ISSB) Scale, and the WHO Quality of Life-BREF (WHOQOL-BREF) Scale.

ELIGIBILITY:
Inclusion Criteria:

* (1) senior residents aged over 60 years, those who were not diagnosed with any cognitive impairment;
* (2) capable of communicating in Mandarin or Taiwanese; and
* (3) capable of using smartphones.

Exclusion Criteria:

* (1) participants who could not fully complete the 8-week intervention (or participate in the course for at least three days per week); and
* (2) those who were incapable of understanding the content of the questionnaire.

Ages: 65 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
UCLA Loneliness Scale (UCLA) | 10-20 minutes
  The third version of UCLA compiled by Russel (1996) was used to measure "loneliness." It was translated into Chinese by Chang and Yang (1999) and included 20 questions. Each question was scored on the 4-point Likert Scale, with 1: "I never feel this way," 2: "I rarely feel this way," 3: "I sometimes feel this way," and 4: "I often feel this way." The total score ranged between 20 and 80, and the higher the score, the higher the participant's degree of loneliness. In this study, the Cronbach's alpha of the pre- and post-intervention UCLA was 0.76 and 0.78, respectively.

SECONDARY OUTCOMES:
Geriatric Depression Scale Short Form (GDS-SF) | 10-20 minutes
  Developed by Sheikh and Yesavage (1986), GDS-SF comprises 15 Yes or No questions, with participants scoring 1 if answering "Yes" or 0 if answering "No." The 2-point scale (Yes/No) made the questionnaire easy to complete for the participants. The threshold of the scale was 7 points, with scores larger than 7 indicating a depression status. The total score ranged between 0 and 15, and the higher the score, the higher the degree of depression. In this study, the Cronbach's alpha of the pre- and post-intervention GDS-SF was 0.81 and 0.82, respectively.
Inventory of Socially Supportive Behavior (ISSB) Scale | 10-20 minutes
  Initially developed by Barrera Jr et al. (1981), ISSB was subsequently translated into Chinese and compiled into 8 questions by Ou (2013). The scale consisted of two categories, namely Emotional Support and Tangible Support. The total score of both categories represented the participant's satisfaction with social support. The scale was scored on a 5-point Likert Scale, with 1 representing "Strongly disagree," 2: "Disagree," 3: "Neutral," 4: "Agree," and 5: "Strongly agree." The total score ranged between 8 and 40, and the higher the score, the higher the participant's satisfaction with social support. In this study, the Cronbach's alpha of the pre- and post-intervention ISSB was 0.83 and 0.77, respectively.
WHO Quality of Life-BREF (WHOQOL-BREF) Scale | 10-20 minutes
  The questionnaire was composed of questions on QOL formulated by the World Health Organization (WHO) based on the commonality of various cultures. The Taiwanese version of WHOQOL-BREF included 28 questions, each scored on a 5-point Likert Scale. It was composed of four domains, namely, Physical health (7 questions), Psychological health (6 questions), Social relationships (4 questions), and Environment (9 questions). The score of an individual question ranged between 1 and 5, and after conversion, the total score of each domain ranged between 4 and 20. The higher the score, the higher the individual's QOL. In this study, the Cronbach's alpha of the domains Physical health, Psychological health, Social relationships, and Environment before and after the intervention was 0.82 (0.80), 0.77 (0.79), 0.76 (0.81), and 0.82 (0.84), respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Asia Univeraity, Taichung, WuFeng, Taiwan